CLINICAL TRIAL: NCT07108101
Title: Interactions Between Placebo Effects and Mindful Awareness State
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 467254
Record Dates: First submitted 2025-05-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Placebo Effect; Mindfulness; Pain; Transcranial Direct Current Stimulation (tDCS)
MeSH Terms: conditions — Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- mindfulness (session 1)+ real tdcs, sham tdcs (session 2) (Experimental): Assigned to the mindfulness group in session 1. Will experience real tdcs, followed by sham tdcs for session 2.
  Interventions: Behavioral: tDCS stimulation (sham); Behavioral: tDCS stimulation (real); Behavioral: Mindful state induction
- mindfulness (session 1) + sham tcds, real tdcs (session 2) (Experimental): Assigned to the mindfulness group in session 1. Will experience sham tdcs, followed by real tdcs for session 2.
  Interventions: Behavioral: tDCS stimulation (sham); Behavioral: tDCS stimulation (real); Behavioral: Mindful state induction
- no mindfulness (session 1) + real tdcs, sham tcds (session 2) (Experimental): Assigned to the no-mindfulness control group in session 1. Will experience real tdcs, followed by sham tdcs for session 2.
  Interventions: Behavioral: tDCS stimulation (sham); Behavioral: tDCS stimulation (real); Behavioral: No minfulness induction
- no mindfulness (session 1) + sham tdcs, real tdcs (session 2) (Experimental): Assigned to the no-mindfulness control group in session 1. Will experience sham tdcs, followed by real tdcs for session 2.
  Interventions: Behavioral: tDCS stimulation (sham); Behavioral: tDCS stimulation (real); Behavioral: No minfulness induction

INTERVENTIONS:
Behavioral: tDCS stimulation (sham) — Participants will receive sham tDCS stimulation in a 20 minute long task.
  Targets will be fitted with the tDCS stimulation electrode cap and instructed that they will receive 20 minutes of tDCS stimulation for the task. Sham tDCS will target the motor cortex at 2mA for 15 sec at the beginning of the session, and then the stimulator will turn off. The participant will then sit for the remaining time of the session with the electrode cap on their heads but turned off and not delivering stimulation.
  All participants will receive sham tDCS stimulation (n=120).
Behavioral: tDCS stimulation (real) — In their second session, participants will receive real tDCS stimulation in a 20 minute long task.
  Targets will be fitted with the tDCS stimulation electrode cap and instructed that they will receive 20 minutes of tDCS stimulation for the task. Real tDCS stimulation will target the motor cortex at 2mA for 20 minutes (full duration of task).
  All participants will receive real tDCS stimulation (n=120).
Behavioral: Mindful state induction — Experimenters trained in high-competence and high-warmth will train Group 1 participants on mindful state induction (n=60). Participants will undergo two stages for this training: 1) pain education to increase beliefs in endogenous brain regulatory capacities; and 2) the Stanford Hypnotic Induction Profile (HIP) test of hypnotizability and hypnotic induction of a relaxed state receptive to suggestion.
  In Stage 1, participants will receive education that pain and affect are processes designed to protect the body from danger, which are transmitted rapidly and automatically to the brain. In Stage 2, participants are (a) seated in an upright, alert posture; and (b) receive suggestions that the ability to attend to and discriminate affective perceptions is achievable and that suppressing attention to the body and focusing on the task will allow them to perform optimally under pressure. Mindful state induction will only be explicitly instructed during session 1 for Group 1 participants.
  Arms: mindfulness (session 1) + sham tcds, real tdcs (session 2); mindfulness (session 1)+ real tdcs, sham tdcs (session 2)
Behavioral: No minfulness induction — Participants in the No-mindfulness group will go through comparable stages but with different instructions. In the first stage, they will receive education about pain and affect as protective processes of the body. In the second stage, they will be seated in an upright, alert posture and receive suggestions to focus on the task and suppress attention to the body.
  Arms: no mindfulness (session 1) + real tdcs, sham tcds (session 2); no mindfulness (session 1) + sham tdcs, real tdcs (session 2)

SUMMARY:
In this experiment,the investigators study the effects of interpersonally induced placebo effects and a mindful awareness induction on negative affect. Specifically, it will be examining the effects of interpersonally induced placebo effects (sham tDCS vs. control) and a mindful awareness induction (mindful state vs. control), as well as their interaction. Each group will undergo fMRI scanning and physiological recording will performing the Multimodal Negative Affect Task (MNAT).

DETAILED DESCRIPTION:
This study aims to investigate the effects of interpersonally induced placebo effects and a mindful awareness induction on negative affect. The study will involve 120 participants recruited from the Dartmouth College community, aged between 18 and 55, with an equal distribution of 60 males and 60 females. Participants will be assigned to the role of "patient" and will undergo fMRI scanning and physiological recording while performing the Multimodal Negative Affect Task (MNAT).

The study design follows a 2 x 2 factorial design, examining the effects of interpersonally induced placebo effects (sham tDCS vs. control) and a mindful awareness induction (mindful state vs. control), as well as their interaction. A follow-up transfer assessment (1 week follow-up, session 2) will be conducted to examine the effects of the mindful state on verum motor tDCS stimulation. The participants will be randomly assigned to either the Mindfulness group or the No-mindfulness group, with 60 participants in each group and two sessions for each participant.

In session 1, participants in the Mindfulness group will undergo a Mindful State Induction procedure aimed at promoting safety, relaxation, and receptivity. This induction procedure consists of two stages. In the first stage, participants will receive education about the brain's connection to and regulation of the body, emphasizing the endogenous brain regulatory capacities. The second stage involves a hypnotic induction of a relaxed state of receptivity using the Stanford Hypnotic Induction Profile (HIP) test of hypnotizability. This stage includes reclining the participant, suggesting that they are always in control, and making somatic suggestions to deepen the receptive state. A guided body scan, derived from mindfulness meditation, will further deepen the induced receptive state.

In contrast, participants in the No-mindfulness group will go through comparable stages but with different instructions. In the first stage, they will receive education about pain and affect as protective processes of the body. In the second stage, they will be seated in an upright, alert posture and receive suggestions to focus on the task and suppress attention to the body.

During the transfer test, conducted in a second fMRI session one week later, we will assess transfer to verum, open-label motor-cortex tDCS in an off-on-off design (both groups), with no explicit mindful state induction. No MRI data will be acquired during tDCS to avoid MR artifacts. We will also assess spontaneous use of strategies, including self-regulation and spontaneous adoption of states of mindful acceptance, and test whether these differ across groups.

The analysis will involve assessing self-report measures, fMRI signatures, and autonomic reactivity to cues and task stimuli, similar to Experiment 1. The analysis will also explore the mediating role of interpersonal response (IPIX scores) and participants' initial responses to placebo.

The researchers plan to control for sex, age, and experimenter effects in all analyses and will test for potential biological sex differences, disaggregating the data if necessary. MRI data will not be acquired during tDCS to avoid artifacts, and the study is not designed to directly compare placebo tDCS with verum tDCS. However, it aims to investigate interpersonal and suggestion-related contributions to open-label treatment responses, providing a foundation for future studies on tDCS and its interactions with placebo effects.

ELIGIBILITY:
* No self-reported current or history of depression, bipolar disorder, or other psychiatric diagnosis
* No self-reported current seizure disorder (i.e., seizure within past 10 years), or history of stroke or other major neurological diagnosis that can cause cognitive impairment
* No self-reported current chronic pain, or acute pain within three months of the study period
* No current migraine disorder (i.e., 15 headache days or more in 1 month)
* No use of central nervous system-effective medication or other medication for neurological/psychiatric treatment
* No self-reported substance abuse within the last six months
* No contraindication to MRI or tDCS (e.g., pregnancy, claustrophobia, pacemakers, ear/cochlear implants, shrapnel injuries, clips, or other ferromagnetic/electrical objects/devices, diagnosed brain abnormality such as tumor, or skin lesions on the scalp.)
* No contraindications for induced pain (e.g., no heart disease, high blood pressure, heart surgery, heart problems of any kind, severe asthma, respiratory problems of any kind, fibromyalgia, Raynaud's Syndrome or Disease, chronic pain, diabetes)
* Participants must be capable of performing experimental tasks (e.g., are able to read), are fluent or native speakers of English
* Participants must be able to tolerate the maximum level of thermal pain stimuli (for thermal stimuli)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report subjective pain experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No pain" and "Most intense pain imaginable". Raw units are on a 0-180 scale.
Subjective fear ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report subjective fear experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No fear" and "Most intense fear imaginable"
Cognitive effort ratings | 3-10 sec post-stimulus throughout testing sessions, with all sessions complete within 1 month
  Participants report cognitive effort experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No effort" and "Most effort imaginable"

SECONDARY OUTCOMES:
Electrodermal autonomic responses to painful heat, fear-related images and cognitive effort. | Peri-stimulus throughout testing sessions, with all sessions complete within 1 month
  Skin conductance (EDA) is recorded continuously throughout test sessions and per-stimulus amplitude of canonical stimulus-locked EDA responses is reported in microsiemens (uS). Higher values indicate a higher EDA response.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Wager, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No